CLINICAL TRIAL: NCT05473858
Title: Comparative Study of the Effect of Diode Laser and Oraverse on Reversing the Effect of Articaine 4% Soft Tissue Anasthesia in Children
Brief Title: Oraverse Versus Laser
Acronym: RCT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: sara nabil (Other)
Responsible Party: Sponsor-Investigator, sara nabil, Lecturer of pediatric dentistry, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AlAzhar
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Reversal of Local Anesthesia in Children
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- laser group (Experimental): Patients will be undergoing anesthesia revision by diode laser
  Interventions: Device: diode laser
- oraverse group (Experimental): Patients will be undergoing anesthesia revision by oraverse
  Interventions: Drug: OraVerse Injectable Product

INTERVENTIONS:
Drug: OraVerse Injectable Product — injection of oraverse,
  Arms: oraverse group
Device: diode laser — patient exposed to diode laser
  Arms: laser group

SUMMARY:
clinically assess the reversal of articaine 4% of two different concentration of vasoconcentration soft-tissue local anesthesia in pediatric dentistry using Diode Laser and Oraverse

DETAILED DESCRIPTION:
Patients will be divided randomly into two groups (20 patients in each group) Group (1): Patients will be undergoing anesthesia revision by diode laser Group (2): Patients will be undergoing anesthesia revision by oraverse. Then each group will be subdivided into 2 subgroups (10 patients each) according to type of local anesthetic agent into:

subgroup 1: Articaine 4% with 1:100000 epinephrin &Subgroup 2: Articaine 4% with 1:200000 epinephrin After 30 min of injection corresponding to approximate time of treatment, the patient in each group will be exposed to the reversal agent which may be diode laser or oraverse.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who need to be treated under anesthesia by injecting mandibular first molar infiltration.
2. Cooperative children aged 6 to 10 years old with the ability to understand and respond to the sensation of soft tissue -

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-09-10 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
reversal of local anasthesia | 30 minute
  patient free of lip numbness

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.sara nabil, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided